CLINICAL TRIAL: NCT02538263
Title: Volume-targeted Versus Pressure-limited Noninvasive Ventilation in Patients With Acute Hypercapnic Respiratory Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Zujin Luo, Attending physician, Beijing Chao Yang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BeijingCYH-ICU-001
Record Dates: First submitted 2015-08-27; First posted 2015-09-02 (Estimated); Last update posted 2019-05-22 (Actual); Status verified 2019-05

CONDITIONS: Acute Hypercapnic Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency

ARMS (2):
- Volume-targeted noninvasive ventilation (Experimental): For Volume-targeted noninvasive ventilation, the target VT was set at 10 ml/kg of ideal body weight, with inspiratory positive airway pressure (IPAP) ranging from 10 cmH2O up to 25 cmH2O.
  Interventions: Device: Volume-targeted noninvasive ventilation
- Pressure-limited noninvasive ventilation (No Intervention): For Pressure-limited noninvasive ventilation, IPAP was initially set at 10 cmH2O, and was adjusted by increments of 1-2 cmH2O according to patients' tolerance (up to 25 cmH2O) to obtain a VT of 8-10 ml/kg of ideal body weight and a respiratory rate (RR) less than 25 breaths/min.

INTERVENTIONS:
Device: Volume-targeted noninvasive ventilation
  Arms: Volume-targeted noninvasive ventilation

SUMMARY:
Volume-targeted noninvasive ventilation (VT-NIV), a hybrid mode that targets a preseted tidal volume (VT) by automated adjustment of pressure support, could guarantee the delivered VT over pressure-limited noninvasive ventilation (PL-NIV) with fixed level pressure support. Whether VT-NIV is more effective in improving gas exchange in patients with acute hypercapnic respiratory failure (AHRF) as compared with PL-NIV remains unclear. Our aim was to verify whether in comparison with PL-NIV, use of VT-NIV was more effective in correcting hypercapnia, hence reducing the need for intubation and improving survival in patients with AHRF.

ELIGIBILITY:
Inclusion Criteria:

* acute hypercapnic respiratory failure (AHRF)
* arterial pH <7.35 and ≥7.25
* PaCO2 >45 mmHg

Exclusion Criteria:

* age <18 years
* excessive amount of respiratory secretions or weak cough
* upper airway obstruction
* recent oral, facial or cranial trauma or surgery
* recent gastric or esophageal surgery
* severe metabolic acidosis; severe abdominal distension
* cardiac or respiratory arrest
* PaO2/FiO2 <150 mmHg
* pneumothorax
* severe ventricular arrhythmia or myocardial ischemia
* severe hemodynamic instability despite fluid repletion and use of vasoactive agents
* active upper gastrointestinal bleeding
* lack of cooperation
* refusal to receive NIV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2013-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
The decrease of arterial partial pressure of carbon dioxide (PaCO2) values from baseline to 6 hours after randomization | 6 hours after randomization
  PaCO2 value at baseline minus PaCO2 value at 6 hours after randomization

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Institute of Respiratory Medicine, Department of respiratory and critical care medicine, Beijing Chao-Yang Hospital Jingxi Campus, Capital Medical University, Beijing, China

REFERENCES:
- [Derived] Cao Z, Luo Z, Hou A, Nie Q, Xie B, An X, Wan Z, Ye X, Xu Y, Chen X, Zhang H, Xu Z, Wang J, An F, Li P, Yu C, Liang Y, Zhang Y, Ma Y. Volume-Targeted Versus Pressure-Limited Noninvasive Ventilation in Subjects With Acute Hypercapnic Respiratory Failure: A Multicenter Randomized Controlled Trial. Respir Care. 2016 Nov;61(11):1440-1450. doi: 10.4187/respcare.04619. Epub 2016 Oct 18. PMID 27794079